CLINICAL TRIAL: NCT05485649
Title: Obstetrical & Neurological Outcomes in Individuals With Epilepsy During Pregnancy
Brief Title: Clinical Outcomes of Pregnant Individuals With Epilepsy - Prospective Study
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Esther Bui, Assistant Professor, MD FRCPC, University Health Network, Toronto
Other Study IDs: 20-5753.2
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: Pregnancy; Neonatal; Obstetrical; Anti-seizure medication
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the pregnancy, delivery, neonatal, and epilepsy outcomes in individuals with epilepsy undergoing pregnancy at the Maternal and Infant Health Programs at the University Health Network - Sinai Health and followed for epilepsy at the Toronto Western Hospital Epilepsy Clinic. In particular, we are interested in the association between following recommended epilepsy management guidelines for pregnant individuals with epilepsy and those aforementioned outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. WWE seen at the Toronto Western Hospital Epilepsy Clinic since June 1st 2022.
2. Pregnant at any point between June 1st 2022 and June 1st 2024 (period of enrolment).
3. Diagnosed with epilepsy as per the International League Against Epilepsy (ILAE) 2014 definition of epilepsy.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant individuals with epilepsy seen at the Toronto Western Hospital Clinic.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of adherence to the 2015 Ontario Task Force management of epilepsy in pregnancy | 2 years
  Describe the frequency of adherence to the 2015 Ontario Task Force management of epilepsy in pregnancy (i.e., AED regimen of WWE, frequency of polytherapy, adherence to serum monitoring of lamotrigine, and folic acid supplementation) and its association with year of pregnancy and type of healthcare provider.

SECONDARY OUTCOMES:
Clinical (neurological, obstetrical, neonatal) outcomes during pregnancy | 1 year
  To determine the association between adherence with the aforementioned guidelines and pregnancy, delivery, neonatal, and neurological outcomes when adjusting for baseline possible confounders.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No